CLINICAL TRIAL: NCT01435447
Title: Fludarabine/Busulfan and Post-infusion Cyclophosphamide as Conditioning for Adult Patients With Lymphoid Malignancies Undergoing Allogeienc Stem Cell Transplantation
Brief Title: Fludarabine/Busulfan and Cyclophosphamide Conditioning for Adult Lymphoid Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Head, Blood and Marrow Transplantation Center, Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJH-ALL-2011
Record Dates: First submitted 2011-09-14; First posted 2011-09-16 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Lymphoid Malignancies
Keywords: efficacy; safety; conditioning; fludarabine; busulfan; cyclophosphamide; adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FLu-Bu-Cy (Experimental): Patients received Fludarabine and iv Busulfan and post-infusion Cyclophosphamide as conditioning
  Interventions: Drug: FLu-Bu-Cy

INTERVENTIONS:
Drug: FLu-Bu-Cy — Fludarabine at 30mg/m2 daily followed by iv-Busulfan at 3.2mg/kg daily for a total of 4 days from Day-6 to -3 and cyclophosphamide as 60mg/kg daily for 2 days on Day +3 and +4, CSA 3mg/kg starting after D+5.
  Other Names: Study group

SUMMARY:
Allogeneic stem cell transplantation is potential curative therapy for adult lymphoid malignancies. Based on our previous study, the condition with iv-busulfan (iv-BU) and cyclophosphamide (CTX) is feasible with low toxicity and transplantation mortality and long-term survival is comparable to most data reported with slightly higher relapse rate particularly for patients in CR2. In this study, the investigators aim to further improve the conditioning with Fludarabine + iv-BU and to use CTX after stem cell transfusion as consolidation for lymphoid malignancies and graft-versus-host disease (GVHD) prophylaxis.

DETAILED DESCRIPTION:
Patients with adult lymphoid malignancies received conditioning with Fludarabine + iv-BU. The GVHD was consisting of D+3 and D+4 CTX after stem cell transfusion. CSA will be added for all patients after D+5.

ELIGIBILITY:
Inclusion Criteria:

* adult acute lymphocytic leukemia in 1st or second remission; lymphoid malignancies in 1st or second remission
* age 16-60 years
* with inform consent
* no contraindication for allogeneic transplantation: active infection, allergy to FLu/Bu/CTX, liver and renal function damage
* HLA matched related (6/6), unrelated donors (at least 8/10) or mismatched related donor (haplo)

Exclusion Criteria:

* age less than 16 years or over 60 years
* liver function/renal function damage (over 2 X upper normal range)
* with mental disease
* other contraindication of all-HSCT

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
acute graft versus host disease (GVHD) | day 100
  d100 incidence of acute GVHD, grade II-IV or grade III-IV
chronic GVHD | 3 years
  3-year incidence of chronic GVHD and extensive cGVHD

SECONDARY OUTCOMES:
non-relapse mortality (NRM) | 3 years
  estimated 3-year NRM after transplantation (death not due to relapse disease)
cumulated incidence of relapse (CIR) | 3 years
  estimated 3-year CIR after transplantation
event-free survival (EFS) | 3 years
  estimated 3-year EFS estimated 3-year EFS after transplantation
overall survival (OS) | 3 years
  estimated 3-year OS after transplantation
GVHD-free, relapse-free survival (GRFS) | 3 years
  estimated 3-year survival for patients without relapse, without III-IV aGVHD and without cGVHD required systemic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Hu, m.D., Principal Investigator — Rui Jin Hospital, Shanghai JiaoTong University School of Medicine
Locations (1):
- Blood and Marrow Transplantation Center, Rui Jin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No